CLINICAL TRIAL: NCT04753866
Title: Facial Scanning for Lip Support Assessment in Full Arch Implant Rehabilitations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implantology Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: II2020-06
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-02

CONDITIONS: Lip; Prosthesis User; Soft Tissue
Keywords: Dental Esthetics; Dental Implants; Three-Dimensional Imaging; Oral Surgery
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia

STUDY DESIGN:
Intervention Model Description: Patients will be quantifiably evaluated regarding facial esthetics and compared before and after the full arch implant supported rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitated (Experimental): Initial lip support condition of the patient when presents himself/herself at the office with indication for full arch implant rehabilitation. Then, the patient is facially scanned before and after the implant surgery.
  Interventions: Device: Facial scanner

INTERVENTIONS:
Device: Facial scanner — The Bellus3D facial scanner will be used to scan the patient before and after implant rehabilitation in order to produce .obj files that allow 3D comparisons and to obtain discrepancy values regarding lip support.

SUMMARY:
Lip support plays an important role in facial esthetics, being a relevant factor when realizing full arch implant supported rehabilitations. However, there is a lack of research on the three dimensional impact of such restorations.

DETAILED DESCRIPTION:
As lip support is becoming more determinant in the facial esthetics outcome after full arch implant rehabilitation, there is a need to know the influence of said rehabilitation in the lower third profile of the patients. Then, through facial scanning, this study's purpose is to evaluate three dimensional changes that arise since the initial state that the patient presents to the office until is rehabilitated through 3D discrepancies and 2D linear measurements.

ELIGIBILITY:
Inclusion Criteria:

* Indication for full arch implant rehabilitation

Exclusion Criteria:

* Presence of facial hair, braces, make up, earrings or any facial deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Lip Support Changes in 3D (μm) | 1 month
  Quantitatively measure 3D facial alterations induced by full arch implant rehabilitation (in Root Mean Square)

SECONDARY OUTCOMES:
Facial Alterations in 2D (mm) | 1 month
  Evaluate facial modifications caused by full arch implant rehabilitation by measuring distances between pre-determined facial landmarks

CONTACTS AND LOCATIONS:
Overall Officials: João Caramês, DDS PhD, Study Director — Implantology Institute; Duarte Marques, DDS PhD, Principal Investigator — Implantology Institute
Locations (1):
- Instituto de Implantologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No